CLINICAL TRIAL: NCT00885001
Title: The Effects of Short Arc Banding: A Novel Exercise Intervention in Patients With Chronic Low Back Pain
Brief Title: The Effects of Short Arc Banding
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Logan College of Chiropractic (Other)
Responsible Party: Dr. Adam Morrell, Logan College of Chiropractic
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RD0311090179; 403
Record Dates: First submitted 2009-04-17; First posted 2009-04-21 (Estimated); Last update posted 2009-04-21 (Estimated); Status verified 2009-04

CONDITIONS: Chronic Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Short Arc Banding Group (Experimental): Lumbar extension on the ATM II from back project. Rehabilitation exercise intervention.
  Interventions: Procedure: Short Arc Banding

INTERVENTIONS:
Procedure: Short Arc Banding — Lumbar extension on the ATM II from back project. Rehabilitation exercise intervention.

SUMMARY:
The general purpose of this pilot study is to determine the effects of a novel exercise intervention (short arc banding (SAB)) on the cross sectional area of lumbar multifidus well as functional outcomes assessments in patients with chronic low back pain.

DETAILED DESCRIPTION:
Multifidus muscle is well known and documented to be a segmental spinal stabilizer and postural muscle. (Bajek, Bogduk) Previous studies have shown evidence that patients with low back pain (LBP) present with multifidus muscle atrophy. It has been documented that patients presenting with unilateral back pain demonstrate an ipsilateral state of reduced cross sectional area of lumbar multifidus (LM) at the segmental level of injury or pain.(Barker, Hides) Chronic LBP sufferers demonstrate a localized and segmentally specific decrease in cross sectional area of multifidus.(Hides) It has been theorized that multifidus muscle surrounding a chronically painful or degenerative segment is less able to stabilize the spine at that segment, predisposing chronic LBP patients to exacerbation due to the inability to cope with demands of day to day life. (Bajek)

Rehabilitative Ultrasound Imaging (RUSI) has been verified as accurate and reliable in determining cross sectional area of lumbar multifidus (Hides). The interrater and intrarater reliability of RUSI has been shown high utilizing a standardized protocol. (Hides) Measurement of LM contraction using RUSI has been shown a valid and useful measure to determine activation of LM as correlated with EMG. (Kiesel) RUSI has been correlated with MRI which is the gold standard for measuring CSA of LM. (Hides)

Type I muscle fibers are the predominant muscle fiber type in lumbar multifidus which has led researchers to pursue spinal stabilization exercises which focus on isometric contractions. These interventions stimulate mainly Type I muscle fibers because they do not use speed or loading parameters theorized necessary to stimulate Type II fibers. (Rissanen, Ng) Previous studies by Rantanen examined LM fiber type in post surgery low backs. Patients with good recovery (minimal to no symptoms 5 years after surgery) showed increased Type II muscle fiber type in relation to those with a poor recovery and Type I fibers increased. (Rantanen) Limited mobility might account for decrease in diameter in Type II fibers in patients undergoing lumbar surgeries.

Notably, Type I muscle fibers appear to increase in size in the presence of chronic LBP. This is probably due to chronic pain induced low tension muscle spasm. (Mattila, Rantanen) Stokes suggested that LM takes on an increasing role in spinal stability due to atrophy of other muscles, thus the increase in size of Type I fibers versus Type II.

To date, the effects of a short arc fast tapping exercise with band resistance or short arc banding (SAB) on the cross sectional area of multifidus has not been documented in the literature. Short arc banding is a novel exercise treatment and to our knowledge is the first study of this mode of exercise. Using a fast motion against band resistance we hope to reach threshold necessary to stimulate not only type I muscle fibers which predominate the LM, but also type II muscle fibers. From the literature, type II muscle fibers decrease in cross sectional area in the presence of a segmental spinal lesion such as lumbar disc herniation. Type II muscle fibers of multifidus aid the spine to respond to and stabilize a ballistic load. Since modern man is much more sedentary, lumbar spines are not loaded adequately to produce stimulation and maintain size of Type II muscle fibers

ELIGIBILITY:
Inclusion Criteria:

* Chronic mechanical low back pain (LBP) with a duration of greater than six weeks, severity and location remaining the same
* No current radicular symptoms extending below the knee
* Logan College Faculty, staff, as well as patients from any of Logan Health Center's allied clinics

Exclusion Criteria:

* Current radicular symptoms extending below the knee
* A history of neurological disease,
* History of severe lumbar trauma or surgery
* Contraindications to lumbar manipulation
* Current use of muscle relaxants or analgesics
* Degenerative joint disease (DJD)
* Recent spinal manipulative therapy (within 2 weeks of start of trial)
* Current use of modalities (e-stim, vibration, etc) and other exercise
* Diabetes
* Heart, kidney thyroid disorders and chronic disease
* Female subjects who are pregnant or breast feeding

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-04; Primary Completion 2009-05 (Estimated); Study Completion 2009-05 (Estimated)

PRIMARY OUTCOMES:
Diagnostic ultrasound | beginning of the trial, at the two week mark and the end of the trial

SECONDARY OUTCOMES:
Revised Oswestery Low Back Disability Questionnaire | at the beginning and end of the trail
Quadruple Visual Analogue Scale | Beginning and end of the trial

CONTACTS AND LOCATIONS:
Locations (1):
- Logan College of Chiropractic, Chesterfield, Missouri, United States